CLINICAL TRIAL: NCT05858138
Title: To Explore the Effectiveness of Jing-Si Herbal Tea Against Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Chun Chiu, Principal Investigator, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REC110-74
Record Dates: First submitted 2023-04-26; First posted 2023-05-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Jing-Si Herbal Tea
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Jing-Si Herbal Tea group (Experimental): Each patient will receive Jing-Si Herbal Tea two times (after breakfast and lunch) in a day for 24 weeks.
  Interventions: Other: Jing-Si Herbal Tea
- Placebo group (Placebo Comparator): Each patient will receive placebo two times (after breakfast and lunch) in a day for 24 weeks.
  Interventions: Other: Placebo Jing-Si Herbal Tea

INTERVENTIONS:
Other: Jing-Si Herbal Tea — patient will receive twice in a day for 24 weeks
  Arms: Jing-Si Herbal Tea group
Other: Placebo Jing-Si Herbal Tea — Placebo Jing-Si Herbal Tea
  Arms: Placebo group

SUMMARY:
The aim of this study is to explore the effectiveness of Jing-Si Herbal Tea on improving the Non-alcoholic fatty liver disease patients

DETAILED DESCRIPTION:
This study adopted a randomized double-blind design, 2-arm trial study. All eligible patients included in the study agreed to participated and signed the informed consent from and the study procedures were approved by the ethical committee of Taichung Tzu Chi general hospital (REC110-74). Patients were recruited from the Gastroenterology department of Taichung Tzu Chi hospital. After random assignment to 2 groups, patients will receive Jing-Si Herbal Tea or placebo twice a day for 24 weeks. We will evaluate the blood test results, abdominal ultrasound and physical examination every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Sign the Informed consent
* Age between 20-70
* Diagnosis for moderated NAFLD
* Liver disease without hepatic decompensation
* HbA1c < = 8.0 %

Exclusion Criteria:

* Do not sign the Informed consent
* Other related liver diseases will affect the study which evaluated by physicians
* Women of potential pregnancy or pregnant women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Assessing the changes from baseline blood glucose at 24 week | 24 week
  Collect the data of blood glucose from blood test
Assessing the changes from baseline GOT (Glutamic Oxaloacetic Transaminase) at 24 week | 24 week
  Collect the data of GOT from blood test
Assessing the changes from baseline GPT (Glutamic Pyruvic Transaminase) at 24 week | 24 week
  Collect the data of GPT from blood test
Assessing the changes from baseline total cholesterol at 24 week | 24 week
  Collect the data of total cholesterol from blood test
Assessing the changes from baseline triglycerides at 24 week | 24 week
  Collect the data of triglycerides from blood test
Assessing the changes from baseline HDL-C at 24 week | 24 week
  Collect the data of HDL-C from blood test
Assessing the changes from baseline LDL-C at 24 week | 24 weekk
  Collect the data of LDL-C from blood test
Assessing the changes from baseline NAFLD activity at 24 week | 24 week
  Scoring the level of NAFLD activity
Assessing the changes from baseline BMI at 24 week | 24 week
  Collect the body height and body weight, weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Tzu Chi Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No